CLINICAL TRIAL: NCT06388668
Title: Timing of Lipid Testing During Hospitalization for MI and Subsequent Management of Dyslipidemia An Observational Study to Reduce the Care Gaps in Dyslipidemia in Canada
Brief Title: Lipid Testing After Myocardial Infarction at the Montreal Heart Institute
Status: Recruiting | Type: Observational
Sponsor: Montreal Heart Institute (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ICM 2025-3428
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-05

CONDITIONS: Dyslipidemias; Lipid Testing; Myocardial Infarction
MeSH Terms: conditions — Dyslipidemias; Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Lipid panel — Lipid panel measuring levels of LDL, non-HDL and apoB

SUMMARY:
Because treatment decisions are usually based on a single measurement of the lipid panel at the time of an admission for an MI, the overarching objective of this project is to evaluate whether the measurement of LDL, non-HDL, and apoB values are reliable through all the duration of the hospitalization.

It will be a single-center, prospective, observational study will be conducted, including consecutive patients hospitalized for myocardial infarction at the Montreal Heart Institute.

Every patient at the Cardiac Care Unit will undergo non-fasting lipid panel testing at day 0 of their admission for Myocardial Infarction during the study period. Patients who consent to participate will have a 2nd non-fasting lipid panel drawn at day 2 of their admission.

Thereafter, the levels of the different lipid values from the panel will be compared between day 0, day 2, and 4-6 weeks after discharge.

DETAILED DESCRIPTION:
We hypothesize that LDL, non-HDL, and apoB values are highest at time of admission and more reflective of the true patient's values, and lower near the time of discharge. Therefore, the timing of testing for the lipid panel during an admission for MI can impact the intensity with which dyslipidemia is treated (i.e. intensity of pharmacologic therapy at discharge), and followed (timing of subsequent lipid panel testing).

The objective of this project is to evaluate whether the measurement of LDL, non-HDL, and apoB values are reliable through all the duration of the hospitalization, from day 0 to day 2.

It will be a single-center, prospective, observational study will be conducted, including consecutive patients hospitalized for myocardial infarction at the Montreal Heart Institute.

Every patient at the Cardiac Care Unit will undergo non-fasting lipid panel testing at day 0 of their admission for Myocardial Infarction during the study period. Patients who consent to participate will have a 2nd non-fasting lipid panel drawn at day 2 of their admission.

The proportion of patients who undergo a repeat lipid panel, and the proportion with a LDL, non-HDL, or apoB value above the intensification threshold, at 4-6 weeks post-discharge, will be assessed. There will be no contact with participants after discharge.

A sample size of 80 to100 patients is aimed for in this exploratory study, based on feasibility and convenience. This sample size is however likely to provide enough power for the primary objective of comparing LDL levels on day 0 and day 2.

Statistical analysis will be conducted at the two-sided 0.05 significance level and performed with SAS.

LDL levels at day 0 and at day 2 will be compared using a paired Student t-test. The changes in LDL from day 0 to day 2 will be estimated and presented with a 95% confidence interval. Results will also be graphically displayed in a bar graph.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18 years old
* Hospitalized at the Cardiac Care Unit for Myocardial Infarction (either NSTEMI or STEMI)
* Lipid panel performed on day 0 of admission
* Willing to provide informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients hospitalized at the Cardiac Care Unit at the Montreal Heart Institute.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Variation in LDL | Day 0 to day 2
  Evaluation of the variation in LDL levels during a hospital admission for myocardial infarction

SECONDARY OUTCOMES:
Variation in non-HDL and apoB | Day 0 to day 2
  Evaluation of the variation in non-HDL and apoB levels during a hospital admission for myocardial infarction
Evaluation of intensification threshold | Day 0 to day 2
  Among the subgroup of patients who are already treated with lipid-lowering therapy at the time of admission, the proportion of patients with a LDL, non-HDL or apoB value above the intensification threshold

OTHER OUTCOMES:
Repeat lipid panel after discharge | 4-6 weeks
  Evaluation of the proportion of patients discharged after myocardial infarction who undergo a repeat lipid panel after discharge
Evaluation of intensification threshold after discharge | 4-6 weeks
  Evaluation of the proportion of patients discharged after MI with a LDL, non-HDL or apoB value above the intensification threshold after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Marquis-Gravel, MD, MSc, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pearson GJ, Thanassoulis G, Anderson TJ, Barry AR, Couture P, Dayan N, Francis GA, Genest J, Gregoire J, Grover SA, Gupta M, Hegele RA, Lau D, Leiter LA, Leung AA, Lonn E, Mancini GBJ, Manjoo P, McPherson R, Ngui D, Piche ME, Poirier P, Sievenpiper J, Stone J, Ward R, Wray W. 2021 Canadian Cardiovascular Society Guidelines for the Management of Dyslipidemia for the Prevention of Cardiovascular Disease in Adults. Can J Cardiol. 2021 Aug;37(8):1129-1150. doi: 10.1016/j.cjca.2021.03.016. Epub 2021 Mar 26. PMID 33781847
- [Background] Sud M, Han L, Koh M, Abdel-Qadir H, Austin PC, Farkouh ME, Godoy LC, Lawler PR, Udell JA, Wijeysundera HC, Ko DT. Low-Density Lipoprotein Cholesterol and Adverse Cardiovascular Events After Percutaneous Coronary Intervention. J Am Coll Cardiol. 2020 Sep 22;76(12):1440-1450. doi: 10.1016/j.jacc.2020.07.033. PMID 32943162
- [Background] Anderson TJ, Gregoire J, Pearson GJ, Barry AR, Couture P, Dawes M, Francis GA, Genest J Jr, Grover S, Gupta M, Hegele RA, Lau DC, Leiter LA, Lonn E, Mancini GB, McPherson R, Ngui D, Poirier P, Sievenpiper JL, Stone JA, Thanassoulis G, Ward R. 2016 Canadian Cardiovascular Society Guidelines for the Management of Dyslipidemia for the Prevention of Cardiovascular Disease in the Adult. Can J Cardiol. 2016 Nov;32(11):1263-1282. doi: 10.1016/j.cjca.2016.07.510. Epub 2016 Jul 25. PMID 27712954
- [Background] Wang WT, Hellkamp A, Doll JA, Thomas L, Navar AM, Fonarow GC, Julien HM, Peterson ED, Wang TY. Lipid Testing and Statin Dosing After Acute Myocardial Infarction. J Am Heart Assoc. 2018 Jan 25;7(3):e006460. doi: 10.1161/JAHA.117.006460. PMID 29371200
- [Background] Gouda P, Welsh RC, Padarath M, Gregoire JC, Hegele RA, Gupta M. Landscape of Lipid Management Following an Acute Coronary Syndrome Event: Survey of Canadian Specialists. CJC Open. 2020 Aug 31;2(6):625-631. doi: 10.1016/j.cjco.2020.08.009. eCollection 2020 Nov. PMID 33305223
- [Background] Elbarouni B, Banihashemi SB, Yan RT, Welsh RC, Kornder JM, Wong GC, Anderson FA, Spencer FA, Grondin FR, Goodman SG, Yan AT; Canadian Global Registry of Acute Coronary Events (GRACE/GRACE(2)) and Canadian Registry of Acute Coronary Events (CANRACE) Investigators. Temporal patterns of lipid testing and statin therapy in acute coronary syndrome patients (from the Canadian GRACE Experience). Am J Cardiol. 2012 May 15;109(10):1418-24. doi: 10.1016/j.amjcard.2012.01.352. Epub 2012 Mar 3. PMID 22381155
- [Background] Sachdeva A, Cannon CP, Deedwania PC, Labresh KA, Smith SC Jr, Dai D, Hernandez A, Fonarow GC. Lipid levels in patients hospitalized with coronary artery disease: an analysis of 136,905 hospitalizations in Get With The Guidelines. Am Heart J. 2009 Jan;157(1):111-117.e2. doi: 10.1016/j.ahj.2008.08.010. Epub 2008 Oct 22. PMID 19081406
- [Background] Pitt B, Loscalzo J, Ycas J, Raichlen JS. Lipid levels after acute coronary syndromes. J Am Coll Cardiol. 2008 Apr 15;51(15):1440-5. doi: 10.1016/j.jacc.2007.11.075. PMID 18402897
- [Background] Rosenson RS. Myocardial injury: the acute phase response and lipoprotein metabolism. J Am Coll Cardiol. 1993 Sep;22(3):933-40. doi: 10.1016/0735-1097(93)90213-k. PMID 7689082